CLINICAL TRIAL: NCT03761303
Title: Investigation of the Efficacy of Repetitive Transcranial Magnetic Stimulation (rTMS) as an add-on Therapy in Patients With Post-stroke Depression (PSD)
Brief Title: rTMS as an add-on Therapy in Patients With Post-stroke Depression
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No eligible patients could be recruited.
Sponsor: BDH-Klinik Hessisch Oldendorf (Other)
Responsible Party: Principal Investigator, Dr. rer. nat. Simone B. Schmidt, Postdoctoral Researcher, BDH-Klinik Hessisch Oldendorf
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: rTMS-PSD
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Post-stroke Depression
Keywords: rTMS; Escitalopram; add-on therapy

STUDY DESIGN:
Intervention Model Description: All patients will receive standard antidepressant therapy with 15 mg escitalopram (Selective Serotonin Reuptake Inhibitor) per day during the study. The dose of escitalopram is increased in all included patients from 5mg/day (day 1-3), over 10mg/day (day 4-6) to 15mg/day (from day 7).
  Patients in the experimental group (active rTMS stimulation) receive active 10 Hz rTMS stimulation over the left dorsolateral prefrontal cortex (DLPFC) over a period of 20 days, seven days a week (20 sessions). The comparison group receives a duration of equal long sham-stimulation.
  For transcranial magnetic stimulation, the Stimulator "PowerMAG Research 100" (Mag & More, Munich, Germany) is used with a cooled double coil (PMD70-pCool).
Who Masked: Participant, Investigator
Masking Description: The randomization of the patients is carried out by a non-medical employee. This co-worker maintains a randomly generated randomization list, indicating to the particular study code (e.g., TMS-PSD-001; TMS-PSD-002), whether to perform an active or sham treatment. The employee pulls a number from an envelope before beginning the intervention of each enrolled patient and then looks at the list to identify the particular group assignment. There will always be randomization packages of ten patients each. Once these are used up, a new list and a new envelope with study codes are prepared.
  In addition, the "real" and the placebo coils are coded before starting studies (eg "A" and "B"). Only the uninvolved employee is the assignment to the real - or placebo coil known. The uninvolved employee randomly assigns the study code containing the information on which coil to use ("A" or "B"). In this way a blinding of performing physician, patient and the evaluating scientist is guaranteed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active rTMS (Active Comparator): Patients in the intervetion group (active rTMS stimulation) receive active 10 Hz rTMS stimulation over the left dorsolateral prefrontal cortex (DLPFC) over a period of 20 days, seven days a week (20 sessions).
  Interventions: Device: active rTMS
- sham rTMS (Sham Comparator): Patients in the control group receive sham rTMS stimulation over the left dorsolateral prefrontal cortex (DLPFC) over a period of 20 days, seven days a week (20 sessions).
  Interventions: Device: sham rTMS

INTERVENTIONS:
Device: active rTMS — The rTMS coil is applied tangentially to the head surface above the left DLPF (corresponding to position F3 of the international 10-20 system). For the stimulation intensity, the motor rest threshold of the patient is determined. The motor rest threshold is defined as the minimum intensity that triggers an EMG response with an amplitude> 50 μV in the first right interosseus dorsalis muscle in at least 5 out of 10 cases. The stimulation intensity within the rTMS therapy is 80 percent of the motor rest threshold. In one session, 1,000 pulses are applied in 10 trains at a frequency of 10 Hz (1 train = 100 pulses in 10 s). Between the individual trains there is an inter-train interval of 28 seconds. The total duration of a session is 5:52 minutes. In total, the patient recieve 20 sessions.
  Arms: active rTMS
Device: sham rTMS — Patients in the intervetion group (active rTMS stimulation) receive active 10 Hz rTMS stimulation over the left dorsolateral prefrontal cortex (DLPFC) over a period of 20 days, seven days a week (20 sessions).
  Arms: sham rTMS

SUMMARY:
About 50% of all stroke patients develop post-stroke depression (PSD). A meta-analysis has shown that rTMS treatment can reduce depressive symptoms in PSD patients. In addition to rTMS alone for the improvement of depression, the question arises as to whether a combination therapy of rTMS plus antidepressant medication can achieve a stronger or longer-term effect in PSD patients. Unfortunately, there are currently no trials of combination therapy with rTMS and drug therapy in PSD patients. Therefore, this study will investigate whether combination therapy of antidepressant and rTMS can provide additional relief of depressive symptoms compared to antidepressant and sham rTMS therapy. It is assumed that the additional active rTMS achieves a faster normalization of affect and drive than with a sham rTMS, so that the patients benefit from neurorehabilitation measures earlier and more sustainably.

DETAILED DESCRIPTION:
Depression is one of the most common forms of mental illness. According to studies by the World Health Organization (WHO), the World Bank and the European Brain Council [1], depression is the leading disease in Europe and Germany since the early 1990s.

Besides drug or psychotherapeutic treatment, repetitive transcranial magnetic stimulation (rTMS) is currently being used as a new non-invasive therapy for depression. The rTMS applies an electromagnetic coil to the patient's head, creating a magnetic field. Impulses emanating from the coil trigger a multitude of reactions at the point of stimulation which, for example, can alter the metabolism, lead to a release of neurotransmitters and a change in gene expression [2-3]. Pulses with a frequency ≤1Hz lead to a reduction of the excitability of the neurons and to an inhibition of cortical activity. In contrast, frequencies ≥5 Hz increase the excitability of neurons and increase cortical activity [4-5].

A large number of studies has already shown that rTMS in depressive patients leads to an improvement in depressive symptoms and has been shown to have an antidepressant effect [6]. In the United States, rTMS has been approved by the Food and Drug Administration (FDA) since 2008 as a treatment for patients with depression who do not respond to antidepressant drug therapy. The FDA recommends a high-frequency (10Hz) rTMS on the left dorsolateral prefrontal cortex (DLPFC) five days a week for four to six weeks [7]. The stimulation of the DLPFC is based on the valence hypothesis that the right hemisphere specializes in the processing of negative emotions and the left hemisphere is specialized in the processing of positive emotions [8] and the DLPFC controls emotional processing [9-10]. Activation of the left DLPFC is therefore associated with the processing of positive emotions [11].

About 50% of all stroke patients develop post-stroke depression (PSD) [12]. A meta-analysis has shown that rTMS treatment can reduce depressive symptoms in PSD patients [13]. In addition to rTMS alone, it is unkown if a combination therapy of rTMS plus antidepressant medication can achieve a stronger or longer-term antidepressive effect in PSD patients. Unfortunately, there are currently no trials of combination therapy with rTMS and drug therapy in PSD patients. Previous studies with depressive patients provide both results that suggest an additional effect of combination therapy [14-19] and results that found no difference between drug-only therapy and combination with rTMS [20-24]. The comparability of the studies is difficult due to the heterogeneity of the study designs. However, it is noticeable that a younger age (<50 years), an intervention duration of rTMS of four weeks, a higher dose of the antidepressant, an inter-train interval (interval between the trains) of <30 seconds and a total number of pulses of <1250 per day, associated with positive effects. However, further studies are needed that address the issue of an additional effect of combination therapy. In addition, a neurological disease was considered to be an exclusion criterion in some of the studies performed [14-15; 20; 23]. It is therefore questionable whether the study results can be transferred to PSD patients.

Therefore, this study will investigate whether combination therapy of antidepressant and rTMS can provide additional relief of depressive symptoms compared to antidepressant and sham rTMS therapy. It is assumed that the additional active rTMS achieves a faster normalization of affect and drive than with a sham rTMS, so that the patients benefit from neurorehabilitation measures earlier and more sustainably.

ELIGIBILITY:
Inclusion Criteria:

* first insult
* Post-stroke Depression (17 item version of the Hamilton Depression Rating Scale [HAM-D]> 18 points)
* capacity to consent

Exclusion Criteria:

* insufficient cardiorespiratory stability
* previous depression or previous use of antidepressants
* pre-stroke psychological illnesses (eg psychosis, bipolar disorder)
* severe cognitive impairment
* aphasia
* lefthanded
* decreased seizure threshold or history of epileptic seizures
* taking medicines that lower the seizure threshold (local anesthetics, cortisone, alcohol, neuroleptics)
* hemorrhages and cerebral edema (e.g., subarachnoid haemorrhage, intracerebral hemorrhage, subdural hematoma, epidural hematoma)
* fresh and healed head wounds near the area to be stimulated
* missing bone cover (relief spread)
* colonization with a germ requiring isolation (e.g., MRSA, 3MRGN, 4MRGN)
* recent myocardial infarction or higher grade cardiac arrhythmias
* contraindications to rTMS: Metallic or magnetic implants containing iron, cobalt or nickel (e.g., pacemakers, brain pacemakers, automatic insulin pumps, electrodes, plates, clips, implanted hearing aids, dental implants, metal endoprostheses, metal parts, or metal fragments in the body).
* pregnancy
* no consent for study participation by the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Changes of Hamilton Depression Rating Scale [HAM-D; 17 Item Version] | For the clinical assessment of the severity of depression, the HAM-D is collected at the following times: day -7; baseline (day 1 before rTMS stimulation); day 2, day 8, day 15 and day 22).
  The primary endpoint is the change in the HAM-D score. A decrease of at least 50% from baseline on day 29 is considered clinically significant. From this, the responder rate is determined.

SECONDARY OUTCOMES:
HAM-D score ≤8 Points | baseline (day 1 before rTMS stimulation); day 22
  A HAM-D score of ≤8 points is considered a decline in depression and is used to record the remission rate. It is expected that the decrease in the HAM-D from baseline (baseline) to the end of the study (day 22) in the active rTMS group is significantly greater than in the sham rTMS group.
HAM-D score (day -baseline) | baseline (day 1 before rTMS stimulation); day 36
  To analyze the long-term effect the HAM-D score will evaluated at day 36 (follow up). It is expected that the decrease in the HAM-D score from baseline to the follow-up (day 36) is significantly greater in the active rTMS group than in the sham rTMS group.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for rehabilitative Research, BDH-Clinic Hessich Oldendorf, Hessisch Oldendorf, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wittchen HU, Jacobi F. Size and burden of mental disorders in Europe--a critical review and appraisal of 27 studies. Eur Neuropsychopharmacol. 2005 Aug;15(4):357-76. doi: 10.1016/j.euroneuro.2005.04.012. PMID 15961293
- [Result] Barker AT, Jalinous R, Freeston IL. Non-invasive magnetic stimulation of human motor cortex. Lancet. 1985 May 11;1(8437):1106-7. doi: 10.1016/s0140-6736(85)92413-4. No abstract available. PMID 2860322
- [Result] Hausmann A, Weis C, Marksteiner J, Hinterhuber H, Humpel C. Chronic repetitive transcranial magnetic stimulation enhances c-fos in the parietal cortex and hippocampus. Brain Res Mol Brain Res. 2000 Mar 29;76(2):355-62. doi: 10.1016/s0169-328x(00)00024-3. PMID 10762712
- [Result] Mitchell PB, Loo CK. Transcranial magnetic stimulation for depression. Aust N Z J Psychiatry. 2006 May;40(5):406-13. doi: 10.1080/j.1440-1614.2006.01816.x. PMID 16683966
- [Result] Milev RV, Giacobbe P, Kennedy SH, Blumberger DM, Daskalakis ZJ, Downar J, Modirrousta M, Patry S, Vila-Rodriguez F, Lam RW, MacQueen GM, Parikh SV, Ravindran AV; CANMAT Depression Work Group. Canadian Network for Mood and Anxiety Treatments (CANMAT) 2016 Clinical Guidelines for the Management of Adults with Major Depressive Disorder: Section 4. Neurostimulation Treatments. Can J Psychiatry. 2016 Sep;61(9):561-75. doi: 10.1177/0706743716660033. Epub 2016 Aug 2. PMID 27486154
- [Result] Schutter DJ. Antidepressant efficacy of high-frequency transcranial magnetic stimulation over the left dorsolateral prefrontal cortex in double-blind sham-controlled designs: a meta-analysis. Psychol Med. 2009 Jan;39(1):65-75. doi: 10.1017/S0033291708003462. Epub 2008 Apr 30. PMID 18447962
- [Result] Horvath JC, Mathews J, Demitrack MA, Pascual-Leone A. The NeuroStar TMS device: conducting the FDA approved protocol for treatment of depression. J Vis Exp. 2010 Nov 12;(45):2345. doi: 10.3791/2345. PMID 21189465
- [Result] Prete G, Laeng B, Fabri M, Foschi N, Tommasi L. Right hemisphere or valence hypothesis, or both? The processing of hybrid faces in the intact and callosotomized brain. Neuropsychologia. 2015 Feb;68:94-106. doi: 10.1016/j.neuropsychologia.2015.01.002. Epub 2015 Jan 7. PMID 25575451
- [Result] Brennan S, McLoughlin DM, O'Connell R, Bogue J, O'Connor S, McHugh C, Glennon M. Anodal transcranial direct current stimulation of the left dorsolateral prefrontal cortex enhances emotion recognition in depressed patients and controls. J Clin Exp Neuropsychol. 2017 May;39(4):384-395. doi: 10.1080/13803395.2016.1230595. Epub 2016 Sep 23. PMID 27662113
- [Result] Zilverstand A, Parvaz MA, Goldstein RZ. Neuroimaging cognitive reappraisal in clinical populations to define neural targets for enhancing emotion regulation. A systematic review. Neuroimage. 2017 May 1;151:105-116. doi: 10.1016/j.neuroimage.2016.06.009. Epub 2016 Jun 8. PMID 27288319
- [Result] Mondino M, Thiffault F, Fecteau S. Does non-invasive brain stimulation applied over the dorsolateral prefrontal cortex non-specifically influence mood and emotional processing in healthy individuals? Front Cell Neurosci. 2015 Oct 14;9:399. doi: 10.3389/fncel.2015.00399. eCollection 2015. PMID 26528131
- [Result] Aben I, Verhey F, Strik J, Lousberg R, Lodder J, Honig A. A comparative study into the one year cumulative incidence of depression after stroke and myocardial infarction. J Neurol Neurosurg Psychiatry. 2003 May;74(5):581-5. doi: 10.1136/jnnp.74.5.581. PMID 12700297
- [Result] Deng L, Sun X, Qiu S, Xiong Y, Li Y, Wang L, Wei Q, Wang D, Liu M. Interventions for management of post-stroke depression: A Bayesian network meta-analysis of 23 randomized controlled trials. Sci Rep. 2017 Nov 28;7(1):16466. doi: 10.1038/s41598-017-16663-0. PMID 29184194
- [Result] Rumi DO, Gattaz WF, Rigonatti SP, Rosa MA, Fregni F, Rosa MO, Mansur C, Myczkowski ML, Moreno RA, Marcolin MA. Transcranial magnetic stimulation accelerates the antidepressant effect of amitriptyline in severe depression: a double-blind placebo-controlled study. Biol Psychiatry. 2005 Jan 15;57(2):162-6. doi: 10.1016/j.biopsych.2004.10.029. PMID 15652875
- [Result] Rossini D, Magri L, Lucca A, Giordani S, Smeraldi E, Zanardi R. Does rTMS hasten the response to escitalopram, sertraline, or venlafaxine in patients with major depressive disorder? A double-blind, randomized, sham-controlled trial. J Clin Psychiatry. 2005 Dec;66(12):1569-75. doi: 10.4088/jcp.v66n1212. PMID 16401159
- [Result] Anderson IM, Delvai NA, Ashim B, Ashim S, Lewin C, Singh V, Sturman D, Strickland PL. Adjunctive fast repetitive transcranial magnetic stimulation in depression. Br J Psychiatry. 2007 Jun;190:533-4. doi: 10.1192/bjp.bp.106.028019. PMID 17541116
- [Result] Bretlau LG, Lunde M, Lindberg L, Unden M, Dissing S, Bech P. Repetitive transcranial magnetic stimulation (rTMS) in combination with escitalopram in patients with treatment-resistant major depression: a double-blind, randomised, sham-controlled trial. Pharmacopsychiatry. 2008 Mar;41(2):41-7. doi: 10.1055/s-2007-993210. PMID 18311683
- [Result] Huang ML, Xu Y, Hu JB, Zhou WH, Wei N, Hu SH, Qi HL, Luo BY. [Repetitive transcranial magnetic stimulation combined with antidepressant medication in treatment of first-episode patients with major depression]. Zhejiang Da Xue Xue Bao Yi Xue Ban. 2011 May;40(3):286-90. doi: 10.3785/j.issn.1008-9292.2011.03.010. Chinese. PMID 21671489
- [Result] Wang YM, Li N, Yang LL, Song M, Shi L, Chen WH, Li SX, Wang XY, Lu L. Randomized controlled trial of repetitive transcranial magnetic stimulation combined with paroxetine for the treatment of patients with first-episode major depressive disorder. Psychiatry Res. 2017 Aug;254:18-23. doi: 10.1016/j.psychres.2017.04.005. Epub 2017 Apr 8. PMID 28441583
- [Result] Garcia-Toro M, Pascual-Leone A, Romera M, Gonzalez A, Mico J, Ibarra O, Arnillas H, Capllonch I, Mayol A, Tormos JM. Prefrontal repetitive transcranial magnetic stimulation as add on treatment in depression. J Neurol Neurosurg Psychiatry. 2001 Oct;71(4):546-8. doi: 10.1136/jnnp.71.4.546. PMID 11561046
- [Result] Hausmann A, Kemmler G, Walpoth M, Mechtcheriakov S, Kramer-Reinstadler K, Lechner T, Walch T, Deisenhammer EA, Kofler M, Rupp CI, Hinterhuber H, Conca A. No benefit derived from repetitive transcranial magnetic stimulation in depression: a prospective, single centre, randomised, double blind, sham controlled "add on" trial. J Neurol Neurosurg Psychiatry. 2004 Feb;75(2):320-2. PMID 14742619
- [Result] Poulet E, Brunelin J, Boeuve C, Lerond J, D'Amato T, Dalery J, Saoud M. Repetitive transcranial magnetic stimulation does not potentiate antidepressant treatment. Eur Psychiatry. 2004 Sep;19(6):382-3. doi: 10.1016/j.eurpsy.2004.06.021. PMID 15363481
- [Result] Herwig U, Fallgatter AJ, Hoppner J, Eschweiler GW, Kron M, Hajak G, Padberg F, Naderi-Heiden A, Abler B, Eichhammer P, Grossheinrich N, Hay B, Kammer T, Langguth B, Laske C, Plewnia C, Richter MM, Schulz M, Unterecker S, Zinke A, Spitzer M, Schonfeldt-Lecuona C. Antidepressant effects of augmentative transcranial magnetic stimulation: randomised multicentre trial. Br J Psychiatry. 2007 Nov;191:441-8. doi: 10.1192/bjp.bp.106.034371. PMID 17978325
- [Result] Huang ML, Luo BY, Hu JB, Wang SS, Zhou WH, Wei N, Hu SH, Xu Y. Repetitive transcranial magnetic stimulation in combination with citalopram in young patients with first-episode major depressive disorder: a double-blind, randomized, sham-controlled trial. Aust N Z J Psychiatry. 2012 Mar;46(3):257-64. doi: 10.1177/0004867411433216. Epub 2012 Jan 5. PMID 22391283